CLINICAL TRIAL: NCT00132873
Title: Long-Term, Open-Label, Multi-Center Extension Trial of Xyrem® (Sodium Oxybate) Oral Solution for the Treatment of Narcolepsy
Brief Title: Trial of Xyrem® (Sodium Oxybate) for the Treatment of Narcolepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Senir Director, Clinical Development - Psychiatry, Jazz Pharmaceuticals, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: OMC-SXB-27
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Cataplexy
MeSH Terms: conditions — Narcolepsy; Cataplexy | interventions — Sodium Oxybate; Solutions

INTERVENTIONS:
Drug: Xyrem (sodium oxybate) oral solution — Xyrem (sodium oxybate) oral solution

SUMMARY:
This is a long-term, open-label, extension of the OMC-SXB-7 trial. Participants from the OMC-SXB-7 open-label trial may be entered without any requirement as to length of participation in that trial.

Approximately 70 patients are expected to participate at up to 6 investigative centers located in Canada. The trial will continue for up to 24 months or until marketing approval, whichever occurs sooner.

DETAILED DESCRIPTION:
This trial will be conducted as a long-term, open-label, extension of the OMC-SXB-7 trial. Participants from the OMC-SXB-7 open-label trial may be entered without any requirement as to length of participation in that trial.

Approximately 70 patients are expected to participate at up to 6 investigative centers located in Canada. The trial will continue for up to 24 months or until marketing approval, whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

* Remained on satisfactory treatment with Xyrem® therapy in the OMC-SXB-7 trial
* Signed and dated an informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brain and Sleep Diagnostic Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xyrem (Sodium Oxybate)
Started | 59
Completed | 50
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 3
Not completed — Planned Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xyrem (Sodium Oxybate)
Number analyzed (Participants) | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 47.6 (15.37)
Gender [Number; unit: participants]
  Female | 41
  Male | 17
Region of Enrollment [Number; unit: participants]
  Canada | 59

OUTCOME MEASURES:

1. Primary Outcome: Adverse Experiences
Description: Number of Subjects with treatment-emergent adverse events.
Time Frame: continuous
Measure: Number; unit: participants
Arm/Group | Xyrem (Sodium Oxybate)
Number analyzed (Participants) | 58
participants | 54

2. Primary Outcome: Vital Signs
Description: Average Respiratory Rate at 1 year.
Time Frame: At 1 year
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Xyrem (Sodium Oxybate)
Number analyzed (Participants) | 49
Breaths per minute | 14.0 (2.40)

ADVERSE EVENTS:
Arm/Group | Xyrem (Sodium Oxybate)
Serious Adverse Events (participants affected / at risk) | 11/58
Other Adverse Events (participants affected / at risk) | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyrem (Sodium Oxybate) (N=58)
Coronary Artery Disease (Cardiac disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cellulitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Enterocolitis Infectious (Infections and infestations) | 1
Obesity (Metabolism and nutrition disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Delusional Disorder, Persecutory Type (Psychiatric disorders) | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xyrem (Sodium Oxybate) (N=58)
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Oedema Peripheral (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 13
Urinary Tract Infection (Infections and infestations) | 11
Influenza (Infections and infestations) | 5
Blood Pressure Increased (Investigations) | 3
Weight Increase (Investigations) | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Sciatica (Nervous system disorders) | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less